CLINICAL TRIAL: NCT00559078
Title: Health-related Quality of Life, Mental Health and Psychotherapeutic Considerations for Women Diagnosed With a Disorder of Sexual Development: Congenital Adrenal Hyperplasia
Brief Title: Qualitative Research on Women With Congenital Adrenal Hyperplasia
Acronym: CAH
Status: Completed | Type: Observational
Sponsor: Lehigh University (Other)
Responsible Party: Matthew Malouf, Lehigh University
Other Study IDs: 1-Malouf
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Adrenal Hyperplasia, Congenital; Psychosexual Development; Sexual Development; Intersex; Qualitative; CAH; Interview; Disorder of Sex Development; Telephone; Quality of Life; Mental Health; Counseling
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Ovotesticular Disorders of Sex Development; Disorders of Sex Development; Psychological Well-Being | interventions — Interviews as Topic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAH: Women diagnosed with CAH (either simple virilizing or salt-losing)
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Hour-long, qualitative, phone interview

SUMMARY:
This qualitative interview-based study will investigate the impact that living with congenital adrenal hyperplasia has for women in the following areas: health-related quality of life (HRQL), psychological health, and health-seeking behaviors.

DETAILED DESCRIPTION:
Congenital Adrenal Hyperplasia is a chronic-illness requiring life-long treatment and is caused by an inherited enzyme deficiency that leads to an overproduction of hormones produced by the adrenal glands, which in turn, masculinizes the female genitalia before birth. While the mechanisms by which CAH influences physiological development are understood, the impact of this hormonal elevation on health-related quality of life (HRQL), psychological health, and health-seeking behaviors is less clear. This study is guided by three research questions: (1) how does CAH influence HRQL domains (physical, functional, emotional and interpersonally), (2) how does CAH influence the mental health of women diagnosed with CAH, and (3) how does CAH influence decisions to seek help from a counselor? Semi-structured qualitative interviews will be conducted with women with CAH. Interviews will be analyzed through the Consensual Qualitative Research (CQR) methodology.

ELIGIBILITY:
Inclusion Criteria:

* 46XX, Females
* Diagnosed by a physician with CAH (either simple-virilizing or salt-losing types)
* Willing to complete a brief demographic questionnaire and participate in an hour long telephone interview

Exclusion Criteria:

* Non-classical or late-onset CAH

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women diagnosed with CAH (either simple-virilizing or salt-losing types) living in the United States
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2007-07; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Telephone interview consisting of approximately 7 open ended questions addressing domains of HRQL, Mental Health and Support | 1 hour

SECONDARY OUTCOMES:
Demographic Questionnaire | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Malouf, BA, Study Director — Lehigh University Counseling Psychology; Arpana G Inman, Principal Investigator — Lehigh University Counseling Psychology
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States